CLINICAL TRIAL: NCT01454518
Title: Effectiveness of Ultrasound Guided Hip Infiltration With Local Anesthetic Solution for Pain Control After Hip Arthroscopy
Brief Title: Local Infiltration Analgesia for Hip Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-08-003
Record Dates: First submitted 2011-10-06; First posted 2011-10-19 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Pain
Keywords: hip arthroscopy; post operative analgesia
MeSH Terms: conditions — Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infiltration of local anesthetic (Experimental): 30 ml of ropivacaine 0.5% infiltrated around lateral anterior and medial aspect of hip joint with ultrasound guidance.
  Interventions: Procedure: Infiltration of local anesthetic
- Normal Saline Injection (Placebo Comparator): injection of 30ml normal saline infiltrated around lateral anterior and medial aspect of hip joint with ultrasound guidance.
  Interventions: Procedure: Normal Saline Injection

INTERVENTIONS:
Procedure: Infiltration of local anesthetic — 30 ml of ropivacaine 0.5% infiltrated around lateral anterior and medial aspect of hip joint with ultrasound guidance.
  Arms: Infiltration of local anesthetic
Procedure: Normal Saline Injection — injection of 30ml normal saline infiltrated around lateral anterior and medial aspect of hip joint with ultrasound guidance.
  Arms: Normal Saline Injection

SUMMARY:
The purpose of this study is to examine if ultrasound guided infiltration of local anesthetic solution around the hip joint will provide effective pain control after hip arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* hip arthroscopy
* ages 18-80

Exclusion Criteria:

* history of neurological disease
* diabetes
* pregnancy
* neuropathy
* chronic narcotic use
* allergy to local anesthetic solution
* inability to give consent or cooperate with the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Post operative opioid consumption. | Within 24 hours after surgery
  Amount in milligrams of opioid consumption post surgery in the recovery room and for a 24 hour period.

SECONDARY OUTCOMES:
Pain scores in recovery room. | Within 24 hours of the surgery
  Mesures of pain score using numeric pain rating scale (0=no pain, 10=worst pain) completed by patient in recovery room and every 6 hours for a 24 hour period after discharge from recovery room.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sinha, M.D., Principal Investigator — Saint Francis Hospital
Locations (1):
- Saint Francis Hospital and Medical Center, Hartford, Connecticut, United States